CLINICAL TRIAL: NCT00319462
Title: Localization of Anatomic Point A in Cervical Cancer Patients
Brief Title: Localization of Point A in Cervical Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mackay Memorial Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MMH-I-S-260
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2007-04-19 (Estimated); Status verified 2006-04

CONDITIONS: Cervical Cancer
Keywords: point A, cervical cancer, radiotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: hemoclip

SUMMARY:
Point A, the major critical point for dose specification of intracavitary brachytherapy, is defined as the crossing of uterine artery and ureter in treatment of cervical cancer. However, the currently advocated systems use hypothetical point A (HPA) to estimate the dosimetry of brachytherapy. This study is to localize anatomic point A (APA) of cervical cancer patients for reference of radiotherapy. We will use laparoscopic clipping technique to localize APA for cervical cancer patients during pelvic and paraaortic lymph node sampling. When these patients are receiving brachytherapy, orthogonal radiographs will be obtained after insertion of tandem and colpostats by using Henschke afterloading applicators.

DETAILED DESCRIPTION:
Radiation therapy (RT), with a relevant integration of external beam radiotherapy (EBRT) and intracavitary brachytherapy (ICBT), is an important part in the treatment of cervical cancer. Even though concurrent chemoradiation therapy (CCRT) improves the control of locoregional recurrence and distant metastasis for locally advanced disease, the role of RT remains important and essential. ICBT is an essential component of RT and has been used to deliver a high localized dose to the primary cervical lesion and adjacent parametria with an attempt to minimize dose to nearby normal tissues. The conventional point-based dose prescription systems have been applied for decades. Incorporation of modern imaging techniques, namely computerized tomography (CT), magnetic resonance imaging (MRI) and positron emission tomography (PET) to ICBT, enable radiation oncologists to individualize treatment volumes but yet, not applicable for routine practice. Point A, since defined by Tod and Meredith in 1938 and revised in 1953, has been widely accepted as a sacrosanct reference point for dose prescription of ICBT. Point A was defined as a point 2 cm above the cervical os and 2 cm apart from os on the line perpendicular to uterine axis. It is a hypothetical point representing the crossover of the ureter and uterine artery, located in the paracervical triangle, and is considered as a critical point for radiation tolerance. This definition of point A provides an easy way to prescribe dose in ICBT and integrate with EBRT. However, its dosimetry according to orthogonal radiographs would depend solely on the applicator geometry but not the individual tumor volume or location. The International Commission on Radiation Units and Measurements (ICRU) report 38 proposed a set of guidelines for uniform reporting. Reporting of the dimensions of reference volumes still depends on the geometry of applied applicator and remains difficult for reporting of ICBT. Thus, point A is still used as a reference point for dose prescription and for correlating the treatment outcome in clinical trials. CCRT has been considered as a standard of care for locally advanced cervical cancer. To further dissect the patient population, which may have a benefit of less morbidity from CCRT, but not radical surgery plus subsequent RT, the sampling of pelvic and paraaortic lymph nodes prior to decision of intended surgery has been utilized by performing laparoscopy or laparotomy for stages IB and IIA. Moreover, this sampling procedure can also provide a pathological proof and delineation of lymph nodes at risk for an important reference of RT field design. During sampling procedures, we observed that the point crossing over the ureter and uterine artery could be visualized and marked by using hemoclips. Therefore, the anatomic position of point A could be visualized on the orthogonal films after closure of abdominal wound. In this study, we attempt to compare the location of and the radiation doses to anatomic point A (APA) and hypothetical point A (HPA) during fractionated ICBT.

ELIGIBILITY:
Inclusion Criteria:

* Female,
* Carvical cancer proven by pathology,
* Indicated for lymph node sampling

Exclusion Criteria:

* Patient refuse lymph node sampling,
* History of allergy to metal materials

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2006-11; Study Completion 2007-04 (Estimated)

PRIMARY OUTCOMES:
Distance difference between anatomiacal and hypothetical point A

SECONDARY OUTCOMES:
Difference from prescribed dose between anatomiacal and hypothetical point A

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Jen Chen, MD,PhD, Principal Investigator — Mackay Memorial Hospital
Locations (1):
- Department of Radiation Oncology, Taipei, Taiwan

REFERENCES:
- [Background] Datta NR. From 'points' to 'profiles' in intracavitary brachytherapy of cervical cancer. Curr Opin Obstet Gynecol. 2005 Feb;17(1):35-41. doi: 10.1097/00001703-200502000-00007. PMID 15711409
- [Background] Datta NR, Basu R, Das KJ, Rajasekar D, Pandey CM, Ayyagari S. Problems in reporting doses and volumes during multiple high-dose-rate intracavitary brachytherapy for carcinoma cervix as per ICRU Report 38: a comparative study using flexible and rigid applicators. Gynecol Oncol. 2003 Nov;91(2):285-92. doi: 10.1016/s0090-8258(03)00506-7. PMID 14599857
- [Derived] Wang KL, Yang YC, Chao KS, Wu MH, Tai HC, Chen TC, Huang MC, Chen JR, Su TH, Chen YJ. Correlation of traditional point a with anatomic location of uterine artery and ureter in cancer of the uterine cervix. Int J Radiat Oncol Biol Phys. 2007 Oct 1;69(2):498-503. doi: 10.1016/j.ijrobp.2007.03.038. PMID 17869664